CLINICAL TRIAL: NCT03992339
Title: An Open-label and Single Arm Study of ATG-010 in Patients With Relapsed/Refractory Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: A Study of Evaluating the Safety and Efficacy of ATG-010 in Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Acronym: SEARCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Antengene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATG-010-DLBCL-001
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Results first posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-04

CONDITIONS: Relapsed/Refractory Diffuse Large B-Cell Lymphoma (DLBCL)
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — selinexor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ATG-010 (Experimental): Enrolled patients will be treated with a fixed dose, 60 mg of ATG-010.
  Interventions: Drug: ATG-010 60 mg, orally, twice weekly, each 4 week (28-day) a cycle

INTERVENTIONS:
Drug: ATG-010 60 mg, orally, twice weekly, each 4 week (28-day) a cycle — Enrolled patients will be treated with a fixed dose, 60 mg of ATG-010, orally, twice weekly, each 4 week (28-day) a cycle.
  Other Names: Selinexor

SUMMARY:
This is an open-label, single arm, and registered study of ATG-010 in Patients with Relapsed/Refractory Diffuse Large B-Cell Lymphoma.

DETAILED DESCRIPTION:
This is an open-label, single arm, and registered study. About 60 patients with relapsed/refractory DLBCL plan to be enrolled in about 10 study sites of the study. It is planned that at least 50% (~30 patients) will have the GCB subtype of DLBCL. Enrolled patients will be treated with a fixed dose, 60 mg of ATG-010, orally, twice weekly, each 4 week (28-day) a cycle. Patients should remain on the study treatment of ATG-010, until either PD or occurrence of unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must provide informed consent form (ICF) prior to the first screening procedure.
2. Age ≥18 years.
3. ECOG performance status of ≤ 2.
4. Patients should have estimated life expectancy of >3 months at study entry.
5. Previously treated, pathologically confirmed de novo DLBCL, or DLBCL transformed from previously diagnosed indolent lymphoma (e.g., follicular lymphoma).
6. Patients must have received at least 2 but no more than 5 previous systemic regimens for the treatment of their de novo or transformed DLBCL.
7. Documented clinical or radiographic evidence of progressive DLBCL prior to dosing.
8. Patients must have measurable disease per the revised criteria for response assessment of lymphoma (Cheson, 2014).
9. Patients must not be eligible for high-dose chemotherapy with autologous stem cell transplantation rescue.

Exclusion Criteria:

1. Patients who are pregnant or lactating.
2. DLBCL with mucosa-associated lymphoid tissue (MALT) lymphoma, composite lymphoma (Hodgkin's lymphoma +NHL), or DLBCL transformed from diseases other than indolent NHL or Richter's.
3. Primary mediastinal (thymic) large B-cell lymphoma.
4. Known central nervous system lymphoma or meningeal involvement.
5. Patients whose most recent systemic anticancer therapy include radiation, chemotherapy, immunotherapy, radio-immunotherapy, or any other anticancer therapy other than glucocorticoids < 6 weeks prior to first dose of study drug.
6. Patients who have not recovered to Grade ≤ 1 clinically significant adverse events, or to their baseline, from their most recent systemic anti-DLBCL therapy.
7. Patients with active graft-versus-host disease after allogeneic stem cell transplantation. At least 4 months must have elapsed since completion of allogeneic stem cell transplantation.
8. Major surgery within 2 weeks of first dose of study treatment of ATG-010.
9. Any life-threatening illness, medical condition or organ system dysfunction which, in the Investigator's opinion, could compromise the patient's safety.
10. Active hepatitis B virus or hepatitis C virus infection.
11. Known human immunodeficiency virus infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bingshan Liu, MD, Study Director — Medical Monitor
Locations (18):
- China (18):
  - Anhui Province Cancer Hospital, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Chongqing Universtity Cancer Hospital, Chongqing, Chongqing Municipality
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Wuhan Union Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Affilate Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin blood research institute, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Cancer Hospital of the University of the Chinese Academy of Sciences, Hangzhou, Zhejiang

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ATG-010
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ATG-010
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (11.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 60
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23.94 (3.089)

OUTCOME MEASURES:

1. Primary Outcome: ORR
Description: ORR is defined as the proportion of patients who achieve either complete response (CR) or partial response (PR) according to the revised criteria for response assessment of lymphoma (2014 Lugano criteria: A complete metabolic response requires Score 1, 2, or 3 with or without a residual mass on 5PS(5-point scale using PET-CT). A PR requires a decrease by more than 50% in the sum of the product of the perpendicular diameters of up to six representative nodes or extranodal lesions.)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | ATG-010
Number analyzed (Participants) | 60
Participants | 13

2. Secondary Outcome: PFS
Description: PFS is defined as the duration from start of selinexor treatment to time of central imaging laboratory determined PD (based on 2014 Lugano criteria: Progressive metabolic disease requires Score 4 or 5 with an increase in intensity of uptake from baseline. Progressive disease by CT criteria only requires an increase in the PPDs of a single node by ≥ 50%.)or death from any cause, whichever occurs first.
Time Frame: 12 months
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | ATG-010
Number analyzed (Participants) | 60
month | 1.87 [1.81 to 2.10]

ADVERSE EVENTS:
Time Frame: From study drug dosed to 30 days after last study drug dose, up to 44 months, SAE was collected from consent, an average of 3.7 year.
Arm/Group | ATG-010
All-Cause Mortality (participants affected / at risk) | 43/60
Serious Adverse Events (participants affected / at risk) | 24/60
Other Adverse Events (participants affected / at risk) | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ATG-010 (N=60)
Platelet count dicreased (Investigations) | 9
Neutrophil count decreased (Investigations) | 3
White blood cell count decreased (Investigations) | 2
Dysphagia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 2
Adynamia (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Cause Death (General disorders) | 1
Pain (General disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
COVID-19 pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Cataract (Eye disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Venous thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ATG-010 (N=60)
Platelet count decreased (Investigations) | 59
White blood cell count decreased (Investigations) | 49
Neutrophil count decreased (Investigations) | 48
Weight decreased (Investigations) | 23
Lymphocyte count decreased (Investigations) | 18
Aspartate aminotransferase increased (Investigations) | 12
Alanine aminotransferase increased (Investigations) | 10
Blood creatinine increased (Investigations) | 10
Blood bilirubin increased (Investigations) | 6
Nausea (Gastrointestinal disorders) | 35
Vomiting (Gastrointestinal disorders) | 20
Diarrhoea (Gastrointestinal disorders) | 19
Constipation (Gastrointestinal disorders) | 15
Anemia (Blood and lymphatic system disorders) | 45
Appetite decreased (Gastrointestinal disorders) | 37
Hyponatraemia (Metabolism and nutrition disorders) | 16
Hypokalaemia (Metabolism and nutrition disorders) | 6
Hyperuricaemia (Metabolism and nutrition disorders) | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 6
Adynamia (General disorders) | 18
Fatigue (General disorders) | 6
Upper respiratory tract infection (Infections and infestations) | 8
Insomnia (Nervous system disorders) | 9
Hypothyroidism (Endocrine disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/39/NCT03992339/Prot_SAP_000.pdf